CLINICAL TRIAL: NCT01171664
Title: A Bi-Center, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group Study Evaluating the Safety and Efficacy of STAHIST in Adult Subjects With a History of Seasonal Allergic Rhinitis
Brief Title: Clinical Trial of STAHIST in Seasonal Allergic Rhinitis (SAR) Subjects
Acronym: STA-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Magna Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 105781-2
Record Dates: First submitted 2010-07-27; First posted 2010-07-28 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2010-09

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: Phase 2; SAR; STAHIST
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo containing no active pharmaceutical ingredients
  Interventions: Drug: Placebo
- STAHIST (Experimental): STAHIST tablet for the symptomatic treatment of Seasonal Allergic Rhinitis
  Interventions: Drug: STAHIST

INTERVENTIONS:
Drug: Placebo — Tablet, one BID
  Arms: Placebo
Drug: STAHIST — STAHIST in tablet form dosed one BID
  Arms: STAHIST

SUMMARY:
To report and compare total symptom scores, nasal symptom scores, post-nasal drip symptom scores, and adverse reactions in and between SAR subjects on active drug and SAR subjects on placebo.

DETAILED DESCRIPTION:
This double-blind, placebo-controlled study will evaluate the efficacy and safety of STAHIST vs. placebo over a 2-week period in 100 study subjects with a history of SAR for at least two years. The study will take place in two sites, Louisville, KY and South Bend, IN. SAR symptoms to be scored and compared include: nasal congestion, rhinorrhea, nasal itching, sneezing, and post-nasal drip.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females of any ethnic group between 18 and 60 years of age.
2. History of moderate to severe SAR for at least two years.
3. Subjects' symptoms resulting from the irritation of sinus, nasal and upper respiratory tract tissues will include the five symptoms that are th focus of this study: nasal congestion, rhinorrhea, nasal itching, sneezing, and post-nasal drip. Subjects must have a TSS baseline score of at least 8 on the S5 Subject Diary.
4. Prior to study drug administration, subjects' good health will be confirmed by medical history and physical examination, including pregnancy test (urine dip) before study inception.
5. Allergic hypersensitivity will be confirmed by the physician or well established patient medical history.
6. Subject's compliance with requisite run-in period for each subject will be confirmed by investigator/designee.

Exclusion Criteria:

1. Pregnancy or lactation.
2. Immunotherapy unless at a stable maintenance dose.
3. Presence of a medical condition that might interfere with treatment evaluation or require a change in therapy including but not limited to high blood pressure or urinary retention problems.
4. Alcohol dependence.
5. Use of any other investigational drug in the previous month.
6. Subjects presenting with asthma requiring corticosteroid treatment.
7. Subjects with multiple drug allergies.
8. Subjects known to have an idiosyncratic reaction to any of the ingredients in IMP (STAHIST).
9. Subject who is participating in any other clinical study.
10. Subject who is unable to meet washout requirements.
11. Subject with clinically significant abnormal vital sign or laboratory value that precludes participation.
12. Subject with any family relationship to the sponsor, investigator, or staff of sponsor or investigator.
13. A URI within 4 weeks of study inception.
14. Subjects taking beta blockers or try-cyclic antidepressants. -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2010-09; Primary Completion 2010-10 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Total Symptom Scores(TSS)reported and compared between the two study arms | Twice daily over the 2 week study period
  TSS includes the sum of nasal congestion, rhinorrhea, nasal itching, sneezing, and post-nasal drip

SECONDARY OUTCOMES:
Adverse events--report and assess | Continuous over the two week study period
  Any/all adverse events will be recorded and scored, reported, evaluated, and results will be clinically and statistically compared between the placebo and active drug arms.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Pollard, MD, Principal Investigator — Family Allergy & Asthma Research Institute
Locations (2):
- United States (2):
  - The South Bend Clinic, South Bend, Indiana
  - Family Allergy & Asthma Research Institute, Louisville, Kentucky